CLINICAL TRIAL: NCT05590104
Title: Effect of Hysteroscopic Isthmocele Repair on IVF Outcome: A Randomized Controlled Trial
Brief Title: Hysteroscopic Isthmocele Repair on IVF Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HealthPlus Fertility Center (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Hamed Elbohoty, Reproductive medicine consultant, HealthPlus Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIROIO
Record Dates: First submitted 2022-10-12; First posted 2022-10-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Reproductive Issues; Cesarean Section; Dehiscence; Intrauterine Disorder

STUDY DESIGN:
Masking Description: The allocated groups will be concealed in serially-numbered sealed opaque envelops that was only opened just after recruitment. Women in any of the groups will receive the allocated treatment after their approval to participate in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysteroscopic CS scar defect repair (Experimental): Patient who is randomized to the hysteroscopic repair of CS scar defect will be prepared to have the surgery postmenstrual.
  The surgery will be under general anasthesia. The participants will be placed in the lithotomy position. The cervix will be visualized using a Sims speculum and grasped using a single-toothed tenaculum, and the cervix, fornix, and vagina will be cleaned.
  Dilatation of the cervix till 7 mm. Introduce the resctoscope through the cervix. The surgical correction of the isthmocele is done by resection of the inferior and superior edges or just the inferior edge of the defect with a resectoscopic loop, using pure cutting current, until reaching the muscular layer. Coagulation of fragile vessels at the base or even entire niche. At the end of procedure, flow and pressure of distending medium can be reduced to ensure adequate haemostasis. After that the patient will be prepared for another euoploid embryo transfer.
  Interventions: Procedure: Hysteroscopic CS scar defect repair
- Expectant management (No Intervention): Patient who is randomized to the expectant management will be prepared for another embryo transfer for euoploid embryo.

INTERVENTIONS:
Procedure: Hysteroscopic CS scar defect repair — Dilatation of the cervix till 7 mm. Introduce the resctoscope through the cervix. The surgical correction of the isthmocele is done by resection of the inferior and superior edges or just the inferior edge of the defect with a resectoscopic loop, using pure cutting current, until reaching the muscular layer. Coagulation of fragile vessels at the base or even entire niche. At the end of procedure, flow and pressure of distending medium can be reduced to ensure adequate haemostasis.
  Arms: Hysteroscopic CS scar defect repair

SUMMARY:
Hysteroscopic Isthmocele repair on IVF outcome It aims to assesse the efficacy of Hysteroscopic CS scar defect repair on the clinical pregnancy rate after embryo transfer.

Patients who were diagnosed with significant caesarean section scar defect and had a previous unsuccessful ongoing pregnancy after embryo transfer of one or more euploid embryo and planning for another trial of one euploid embryo transfer will be assed for study eligibility. Twenty five of them will be be randomized to hysteroscopic repair before having embryo transfer. and 25 will go directly for embryo transfer. Clinical pregnancy rate is the primary outcome.

DETAILED DESCRIPTION:
Hysteroscopic Isthmocele repair on IVF outcome Background: Uterine niche is a very common finding in women with previous caesarean section. Subfertility can be associated finding and IVF outcome can be affected by its presence. It is not yet if its treatment before IVF trial could improve the outcome of IVF cycle.

Objectives: assesse the efficacy of Hysteroscopic CS scar defect repair on the clinical pregnancy rate after embryo transfer.

Methods This prospective randomized controled will be conducted at Healthplus fertility center. The population of the study will be Patients who was diagnosed with significant caesarean section scar defect and had a previous unsuccessful ongoing pregnancy after embryo transfer of one or more euploid embryo and planning for another trial of one euploid embryo transfer. Twenty five of them will be be randomized to hysteroscopic repair before having embryo transfer. and 25 will go directly for embryo transfer. Clinical pregnancy rate is the primary outcome. Seconday outcomes are Complications following hysteroscopic CS scar repair, the need of aspiration of intrauterine fluid before embryo transfer, early pregnancy complications, Caesarean section scar dehiscence or rupture and live birth rate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed CS scar defect by TVUS
* At least one failed trial of euploid embryo transfer
* Planning for a trial of single euploid embryo transfer

Exclusion Criteria:

* Residual myometrial thickness less than 3 mm
* Any congenital uterine abnormalities.,
* Prescence of intrauterine lesions e.g. polyp, fibroid, Endometriosis or adenomyosis, Hydrosalpinx, Chronic endometritis, Previous CS scar defect repair.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-03-26 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinical pregnancy | at 7 weeks of gestation or beyond
  detection of intrauterine pregnancy with a detectable fetal heart pulsation by transvaginal ultrasound scan

SECONDARY OUTCOMES:
Rate of Complications following hysteroscopic CS scar repair | up to 6 weeks
  uterine perforation, fluid overload and endometritis
Rate of Need of aspiration of intrauterine fluid | During the preparation of embryo transfer. Through study completion, an average of 1 year
  Presence intrauterine fluid collection at the time of embryo transfer which should be aspirated before embryo transfer
Rate of Early pregnancy complications | 12 weeks gestation
  Ectopic pregnancy or Miscarriage
Rate of Caesarean section scar dehiscence or rupture | Within 40 weeks of pregnancy
  Rupture of CS scar during the antenatal period or presence of CS scar wound dehiscence at the time of delivery
Rate of delivery of a living baby | Within 40 weeks of pregnancy
  Delivery of a living baby after 24 weeks gestation

CONTACTS AND LOCATIONS:
Locations (2):
- United Arab Emirates (2):
  - Healthplus fertility center, Abu Dhabi, UAE
  - Healthplus fertility center, Abu Dhabi

IPD SHARING:
Plan to Share IPD: Yes
This prospective randomized controlled will be conducted at Healthplus fertility center. The population of the study will be Patients who was diagnosed with significant caesarean section scar defect and had a previous unsuccessful ongoing pregnancy after embryo transfer of one or more euploid embryo and planning for another trial of one euploid embryo transfer. Twenty five of them will be be randomized to hysteroscopic repair before having embryo transfer. and 25 will go directly for embryo transfer. Clinical pregnancy rate is the primary outcome. Secondary outcomes are Complications following hysteroscopic CS scar repair, the need of aspiration of intrauterine fluid before embryo transfer, early pregnancy complications, Caesarean section scar dehiscence or rupture and live birth rate.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18 months
Access Criteria: open